CLINICAL TRIAL: NCT01517386
Title: Optical Tissue Stylet (OTS) - Descriptive Observational Study Into Paravertebral Space (PS) Detection in Humans
Brief Title: Photonic Needle and Paravertebral Space Detection
Acronym: OTS-PS
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL37671.091.11
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-07

CONDITIONS: Anesthesia
Keywords: paravertebral space; needle placement; tissue identification; regional
MeSH Terms: interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- paravertebral anesthesia: patients scheduled for elective unilateral thoracic surgery under paravertebral block and general anesthesia
  Interventions: Procedure: thoracic surgery

INTERVENTIONS:
Procedure: thoracic surgery — unilateral thoracic surgery under paravertebral block and general anesthesia

SUMMARY:
For effective anesthesia and interventional pain treatments, correct needle placement is crucial. Currently used methods to guide needle placement and confirm the actual treatment location before injection of the medication include: image-guidance, loss-of-resistance, and electrical stimulation. However, accuracy of needle placement could be improved if information would be available that would complement the current methods. We have developed the so-called "photonic needle" technology based on optical spectroscopy that has the potential to provide such complementary information.

This study is an observational study in a limited number of patients. A common ultrasound-guided regional anesthesia procedure has been selected, during which data will be acquired with the photonic needles at a number of points along the needle trajectory that allow for confirmation by imaging.

Rationale for this study is to investigate the potential of the technology to discriminate tissues that are relevant to distinguish during the procedure.

DETAILED DESCRIPTION:
The primary objective of the trial is to investigate if the photonic needle technology can reliably identify the thoracic paravertebral space. Diffuse reflectance spectra will be acquired during needle advancement, with custom-made needle stylets that contain optical fibers.

Main study parameters are:

1. Successfully acquired diffuse reflectance spectra obtained in the thoracic paravertebral space, and spectra obtained during needle advancement.
2. Confirmation of sonographic thoracic paravertebral localization, defined as tissue imaging in all locations of the needle where the diffuse reflectance spectra have been collected .
3. Recordings of reaction to a small test dose of lidocaine 2% with epinephrine 1:200.000 at target position for regional anesthesia (to exclude vascular localization of the needle)
4. "certainty score" on a 3-point scale (1 = uncertain, 2 = certain, 3 = very certain) provided by the physician for assignment of the type of tissue present at the needle tip, based on the information available from imaging and/or aspiration and/or reaction to a small injection of epinephrineOther study parameters

The endpoint of the study is a statistical analysis of the difference between diffuse reflectance spectra obtained at non-paravertebral and paravertebral measurement locations.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral thoracic surgery
* Age between 18 and 80 years of age
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Pregnancy
* Photodynamic therapy
* Contraindications to regional anesthesia and/or allergy to amide local anesthetics.
* Subjects < 18 years of age or >80 years of age
* Severe coagulopathy
* Subjects with severe thoracic deformities
* Subjects with contraindications to methylene blue

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective unilateral thoracic surgery under paravertebral block and general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Identification of the thoracic paravertebral space | Day 0
  Statistical analysis of the difference between diffuse reflectance spectra obtained at non-paravertebral and paravertebral measurement locations

CONTACTS AND LOCATIONS:
Overall Officials: Gert-Jan Scheffer, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands